CLINICAL TRIAL: NCT05675397
Title: Supplementation of Mother's Own Milk With Preterm Donor Human Milk: Impact on Morbidity and Growth in Very Low Birth Weight Infants
Brief Title: Preterm Donor Human Milk Supplementation of Mother's Own Milk in VLBW Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Soultana (Tania) Siahanidou, Professor in Pediatrics-Neonatology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 6116
Record Dates: First submitted 2022-12-14; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Prematurity
Keywords: preterm infants; nutrition; donor milk; breast milk
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOM supplemented with PDM (group A) (Experimental): VLBW Infants fed with mother's own milk (MOM) supplemented with preterm donor milk (PDM)
  Interventions: Dietary Supplement: donor human milk
- MOM supplemented with TDM (group B) (Active Comparator): VLBW infants fed with mother's own milk (MOM) supplemented with term donor milk (TDM)
  Interventions: Dietary Supplement: donor human milk

INTERVENTIONS:
Dietary Supplement: donor human milk — Pasteurized preterm donor milk (PDM) versus term donor milk (TDM) will be provided to the study population following randomization, as supplementary to mother's own milk (MOM) or as alternative feeding

SUMMARY:
This prospective randomized controlled trial aims to investigate whether feeding very low birth weight (VLBW) infants with Mother's own milk (MOM) supplemented with either preterm (PDM) or term donor milk (TDM), when MOM is insufficient, has a positive impact on infants' protein intake, growth and morbidity.

DETAILED DESCRIPTION:
Mother's own milk (MOM) is the optimal nutrition for preterm infants. When MOM is not sufficient, pasteurized donor milk (DM) is the best alternative according to current recommendations. Donor milk is primarily derived from mothers of term-born infants for the first six months of lactation. However, this term milk presents significant differences compared to preterm human milk which has higher protein concentration and more caloric energy.

The investigators hypothesized that feeding VLBW infants with preterm donor milk (PDM) in combination with MOM may positively influence the protein intake and, consequently, the infants' growth. The aim of the current study is to assess whether MOM supplementation with PDM has any beneficial effects on the nutrition, growth and morbidity in VLBW infants.

ELIGIBILITY:
Inclusion Criteria:

• VLBW infants with birth weight <1500g born to mothers who agree to provide donor milk for the first three weeks of life (donor milk period) if their own milk quantity is insufficient

Exclusion Criteria:

* Congenital anomalies
* Chromosomal disorders
* Metabolic diseases
* Feeding with formula at any point during the first 3 weeks of life (donor milk period)

Ages: 1 Day to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of infants' growth | From randomization to discharge, up to 40 weeks of postconceptional age (term equivalent age)
  Infants' weight gain during hospitalization (grams per day) will be assessed and compared between group A and group B.
Assessment of protein intake | From randomization to discharge, up to 40 weeks of postconceptional age (term equivalent age)
  Protein intake by the study participants during hospitalization (grams per Kg of body weight per day) will be assessed and compared between group A and group B.
Assessment of morbidity | From randomization to discharge, up to 40 weeks of postconceptional age (term equivalent age)
  Culture positive sepsis in study participants during hospitalization will be assessed and compared between group A and group B.

CONTACTS AND LOCATIONS:
Overall Officials: George Liosis, MD, PhD, Study Chair — Neonatal Intensive Care Unit, "Elena Venizelou" General and Maternal Hospital, Athens, 11521, Greece; Giannoula Gialeli, Principal Investigator — Neonatal Intensive Care Unit, "Elena Venizelou" General and Maternal Hospital, Athens, 11521, Greece; Tania Siahanidou, Study Director — First Department of Pediatrics, School of Medicine, National and Kapodistrian University of Athens
Locations (2):
- Greece (2):
  - Neonatal Intensive Care Unit, "Elena Venizelou" General and Maternal Hospital, Athens
  - First Department of Pediatrics, National and Kapodistrian University of Athens, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gialeli G, Kapetanaki A, Panagopoulou O, Vourna P, Michos A, Kanaka-Gantenbein C, Liosis G, Siahanidou T. Supplementation of Mother's Own Milk with Preterm Donor Human Milk: Impact on Protein Intake and Growth in Very Low Birth Weight Infants-A Randomized Controlled Study. Nutrients. 2023 Jan 21;15(3):566. doi: 10.3390/nu15030566. PMID 36771273